CLINICAL TRIAL: NCT05073913
Title: Vascular Remodeling After Living Kidney Donation
Brief Title: Vascular Remodeling After Living Kidney Donation Study
Acronym: EUGENIA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP191038; IDRCB 2020-A00723-36 (Other: ANSM)
Record Dates: First submitted 2021-05-10; First posted 2021-10-12 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Living Kidney Donation
Keywords: living kidney donors; endothelial function; vascular remodeling; pulse wave velocity; glomerular filtration rate
MeSH Terms: conditions — Vascular Remodeling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Living kidney donors (Active Comparator): complete vascular exploration before and one year after nephrectomy
  Interventions: Diagnostic Test: Vascular remodeling characterization
- potential living kidney donors (Sham Comparator): complete vascular exploration before and one year after the first exploration (for patients with medical contraindication to donation or who have declined donation after the first exploration)
  Interventions: Diagnostic Test: Vascular remodeling characterization

INTERVENTIONS:
Diagnostic Test: Vascular remodeling characterization — Pulse wave velocity measure High frequency ultrasonography for vascular imaging Endothelial function test Left ventricular mass by echocardiography Measurement of GFR (Glomerular Filtration Rate) with decrease in plasma of Iohexol

SUMMARY:
Vascular evaluation of candidates to living kidney donation is important because there is an increased risk of end stage renal disease and cardiovascular disease after donation. The implication of vascular remodeling in the vascular morbidity observed in donors has not been established because the parameters of vascular remodeling in donors have so far been poorly described. The object of the present study is to study the evolution of vascular remodeling of small, medium and large vessels (until then not evaluable by standard techniques) before and one year after living kidney donation, by dedicated-, non invasive-examinations, which results are associated with cardiovascular risk in the general population. This approach will make it possible to precisely assess the impact of unilateral nephrectomy on vascular remodeling after living donation and to estimate the change in cardiovascular risk attributable to the donation. These results will also help refine the assessment of candidates for kidney donation and potentially open up new strategies to improve selection process of candidates to living kidney donation. Of note, we also plan to evaluate one year after the first exploration potentiel living kidney donors who did not give their kidney due to medical or non medical reasons, as a control group.

ELIGIBILITY:
Inclusion Criteria:

* candidate to living kidney donation
* affiliated to national health insurance
* capable of understanding the consequences of participating to the study
* written informed consent

Exclusion Criteria:

* pregnancy
* breastfeeding
* allergy to iodinated contrast agents
* allergy to echographic gel, allergy to cutaneous dressings
* cutaneous lesions preventing the ultrasonography probe to be applied on the skin
* participation to a drug trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-05-10 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Carotid artery rigidity | 1 year after living kidney donation or after the first exploration for the non donors
  Carotid stiffness, as measured by echotracking

SECONDARY OUTCOMES:
Measured glomerular filtration rate | 1 year after living kidney donation or after the first exploration for the non donors
Pulse wave velocity | 1 year after living kidney donation or after the first exploration for the non donors
Endothelial function | 1 year after living kidney donation or after the first exploration for the non donors
  Measured Glomerular Filtration Rate (urinary clearance of 99mTc-DTPA) unit: ml/min/1,73 m²
Small arteries remodeling | 1 year after living kidney donation or after the first exploration for the non donors

CONTACTS AND LOCATIONS:
Overall Officials: Marie COURBEBAISSE, MD, PhD, Principal Investigator — marie.courbebaisse@aphp.fr
Locations (1):
- Hôpital Necker, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on scientific project and scientific involvement of the PI team. Collaboration will be fostered. The founder could be involved in the decision.
  Data sharing must respect the agreements made with funders. Teams wishing obtain IPD must meet the sponsor and IP team to present scientific (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractual agreement. contractualization.
  Processing of shared data must comply with European General Data Protection Regulation (GDPR).